CLINICAL TRIAL: NCT05284097
Title: A Phase 2, Open-label, Study to Evaluate the Safety and Immunogenicity of a Heterologous 2-dose Vaccination Regimen Using Ad26.ZEBOV, MVA-BN-Filo in Adults and Children Originally Enrolled in the Control Arm of the EBOVAC-Salone Study
Brief Title: Ad26.ZEBOV, MVA-BN-Filo Vaccination in Children and Adults Previously Vaccinated With Control in the EBOVAC-Salone Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Sierra Leone (Other); Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VAC52150EBL2012
Record Dates: First submitted 2022-02-23; First posted 2022-03-17 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Virus Diseases; Hemorrhagic Fever, Ebola; Infections; Hemorrhagic Fevers, Viral; RNA Virus Infections; Filoviridae Infections; Mononegavirales Infections; Vaccines; Immunologic Factors; Physiological Effects of Drugs; Ebola
Keywords: Ad26.ZEBOV; MVA-BN-Filo; vaccination; children; adults
MeSH Terms: conditions — Virus Diseases; Hemorrhagic Fever, Ebola; Infections; Hemorrhagic Fevers, Viral; RNA Virus Infections; Filoviridae Infections; Mononegavirales Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Intervention (Experimental): Subjects will receive the following study vaccines as a 0.5 mL IM injection into the deltoid:
  * Ad26.ZEBOV at a dose of 5x10^10 vp on Day 1
  * MVA-BN-Filo at a dose of 1x10^8 Inf U on Day 57
  Interventions: Drug: Ad26.ZEBOV, MVA-BN-Filo

INTERVENTIONS:
Drug: Ad26.ZEBOV, MVA-BN-Filo — Ad26.ZEBOV - is an adenovirus serotype 26 vector expressing the glycoprotein (GP) of the Ebola virus (EBOV) Mayinga variant
  MVA-BN-Filo - is a Modified Vaccinia Ankara (MVA) - Bavarian Nordic (BN) vector expressing the GPs of EBOV, Sudan virus (SUDV) and Marburg virus (MARV) and the nucleoprotein of Tai Forest virus
  Other Names: VAC52150

SUMMARY:
This is a Phase 2, open-label, study evaluating the safety and immunogenicity of the 2-dose vaccination regimen, Ad26.ZEBOV, MVA-BN-Filo, in adults and children originally enrolled in the control arm of the EBOVAC-Salone study

DETAILED DESCRIPTION:
This study is being conducted to assess the safety and immunogenicity of the Ad26.ZEBOV (Dose 1), MVA-BN-Filo (Dose 2) vaccine regimen, administered with a 56-day interval between the two doses, in adults and children previously enrolled in the control arm of the VAC52150EBL3001 (EBOVAC-Salone) study.

The heterologous, 2-dose Ebola vaccine regimen is comprised of the following 2 Ebola vaccines:

* Ad26.ZEBOV - an adenovirus serotype 26 vector expressing the glycoprotein (GP) of the Ebola virus (EBOV) Mayinga variant
* MVA-BN-Filo - a Modified Vaccinia Ankara (MVA) - Bavarian Nordic (BN) vector expressing the GPs of EBOV, Sudan virus (SUDV) and Marburg virus (MARV) and the nucleoprotein of Tai Forest virus

STUDY OBJECTIVES AND HYPOTHESIS

Primary Objectives:

* To assess the safety of the Ad26.ZEBOV, MVA-BN-Filo Ebola vaccine regimen administered intramuscularly with a 56-day interval between the two doses.
* To quantify and characterise cellular immune responses to EBOV-GP induced by the Ad26.ZEBOV, MVA-BN-Filo Ebola vaccine regimen as measured by cell mediated immunity assays at 56 days post Dose 1 and 21 days post Dose 2.

Secondary Objective:

• To evaluate humoral immune responses against EBOV GP induced by the Ad26.ZEBOV, MVA-BN-Filo Ebola vaccine regimen as measured by enzyme-linked immunosorbent assay (ELISA) at 56 days post Dose 1 and 21 days post Dose 2.

Exploratory Objectives:

• To characterise binding antibodies induced by the Ad26.ZEBOV, MVA-BN-Filo Ebola vaccine regimen using LUMINEX technology.

Hypothesis:

As this study is designed to provide descriptive information regarding safety and immunogenicity without formal treatment comparisons, no formal statistical hypothesis testing is planned.

OVERVIEW OF STUDY DESIGN This is a Phase 2, open-label study to evaluate the safety and immunogenicity of Ad26.ZEBOV (first vaccination) at a dose of 5x10^10 viral particles (vp) followed by MVA-BN-Filo (second vaccination) at a dose of 1x10^8 infectious units (Inf U) administered 56 days later in healthy adults and children.

Only subjects from the feeder study, VAC52150EBL3001 (EBOVAC-Salone), who were enrolled in the control arm (did not received the Ebola vaccine regimen) are eligible for enrollment in this study.

Potential participants or parents/guardians of potential participants will be asked to consent for their participation or their children's participation in the study. Children aged 7 years and older at the time of enrollment in this study will be asked to give positive assent for their participation. Participants will be followed up for 28 days following Dose 2 vaccination. The study will be conducted in Kambia, Sierra Leone.

Study population: subjects must be healthy adults and children (based on physical examination, medical history, and clinical judgment) who were in the control arm in the VAC52150EBL3001 (also known as EBOVAC-Salone) vaccine trial.

Dosage and administration: subjects will receive the following study vaccines as a 0.5 millilitres (mL) intramuscular (IM) injection into the deltoid:

* Ad26.ZEBOV at a dose of 5x1010 vp on Day 1
* MVA-BN-Filo at a dose of 1x108 Inf U on Day 57

Safety evaluations: for children ages 4-11 years, solicited local (at the injection site) and systemic adverse events will be assessed using a symptom diary for a period of seven days following each vaccination. For all participants, serious adverse events will be reported from Dose 1 vaccination until their last study visit.

Immunogenicity evaluations: blood will be drawn for assessments of humoral and cellular immune responses at the Day 1, Day 57, and Day 78 visits. Blood samples for cellular immune responses will only be collected in a subset of participants; 30 participants aged 4-11 years, 30 participants aged12-17 years, and 30 participants aged 18 years and older.

STATISTICAL METHODS The primary analysis will be conducted when all subjects have completed the 28 days post-Dose 2 visit or discontinued earlier. This analysis will include all available data up to this point.

Sample size determination: up to 245 adults and children will be invited to enroll into this trial and included in safety and humoral immunogenicity evaluations. This number is based on the potentially available participants in EBOVAC-Salone who were enrolled into the control groups.

A randomly selected subset of 90 participants (including 30 aged 4-11 years, 30 aged 12-17 years and 30 aged 18 years and older) will be included in the cellular immunogenicity subset. Inclusion of 90 participants will enable estimation of the proportion of participants with detectable post-vaccination EBOV-specific T cell subsets of interest with an acceptable level of precision.

Safety analysis: no formal statistical testing of safety data is planned. Safety data will be analysed descriptively by age the participant is when s/he received Dose 1 of the Ebola vaccine regimen (Ad26.ZEBOV, MVA-BN-Filo), based on the age groups: 4-11 years, 12-17 years, 18 years and older.

Immunogenicity analyses:

The investigators will calculate the proportion of participants with detectable EBOV-specific T cell subsets of interest at baseline, 56 days post dose 1 and at 21 days post dose 2 with exact binomial 95% confidence intervals (CIs).

A similar approach will be taken in analyses of antibody responses (using both ELISA and LUMINEX). The proportion of participants with an EBOV-specific antibody response will be calculated with 95% CIs at baseline and follow up visits, and the magnitude of the observed antibody responses will be described at each visit using measures of central tendency and spread.

Immunogenicity analyses will be performed first among all participants with contributing data (up to n=245 for humoral responses; n=90 for cellular responses), and second stratified by age group.

ELIGIBILITY:
Inclusion Criteria:

1. Must have been enrolled in the control arm and received at least the first vaccination (Dose 1) in EBOVAC-Salone.
2. Must consent to participate, or their parent/guardian must consent for their child to participate, in the VAC52150EBL2012 study.Children aged 7 years and older will be asked to give positive assent for their participation in the study.
3. Must be willing/able to adhere to the prohibitions and restrictions specified in the protocol, or the parent/guardian must be willing/able to ensure that their child adheres to the prohibitions and restrictions specified in the protocol
4. Must be healthy in the investigator's clinical judgement (and the parent/guardian's judgement) on the basis of medical history, physical examination, vital signs, and a haematological assessment (i.e., full blood count) performed at screening.
5. Female subjects of childbearing potential, who have started their menstrual periods and/or are ≥12 years of age at the time of screening must use adequate birth control measures consistent with local regulations regarding the use of birth control for subjects participating in clinical studies from at least 14 days before vaccination until the end of the study, with a negative urine beta human chorionic gonadotropin (β-hCG) pregnancy test at screening and immediately prior to the vaccination, which shall occur no earlier than 14 days after the screening visit.
6. Must be willing to participate for the duration of the study visits, or the parent/guardian must be available and willing to have their child participate for the duration of the study visits.
7. Must have, or the parent/guardian must have, the means to be contacted.
8. Must pass the Test of Understanding (TOU), or the parent/guardian must pass the TOU.

Exclusion Criteria:

1. Participants in the EBOVAC-Salone trial who received at least 1 dose of the Ebola vaccine regimen.
2. Subjects who have received any candidate or other Ebola vaccine.
3. Subjects who have a known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccine, e.g., polysorbate 80, ethylenediaminetetraacetic acid, or L-histidine for Ad26.ZEBOV vaccine), including known allergy to chicken or egg proteins and aminoglycosides (gentamicin).
4. Subjects who have a known history of any thrombotic disorder, thrombocytopaenia, thrombotic thrombocytopaenia syndrome (TTS), or heparin-induced thrombocytopaenia and thrombosis (HITT).
5. Subjects with presence of acute illness (this does not include minor illnesses such as mild diarrhoea or mild upper respiratory tract infection) or axillary temperature ≥38° C on Day 1. Participants with such symptoms will be excluded from enrolment at that time but may be rescheduled for enrolment at a later date within the screening window.
6. Subjects with a clinically significant history of skin disorder (e.g., psoriasis, contact dermatitis), allergy, symptomatic immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness as judged by the investigator or other delegated individual.
7. Women who are known to be pregnant or planning to become pregnant while enrolled in the study.
8. Subjects who have received a blood transfusion or other blood products within 8 weeks prior to vaccination day.
9. Subjects who have been vaccinated with live-attenuated vaccines within 30 days before the study vaccination, or with an inactivated vaccine within 15 days before the study vaccination.
10. Subjects who, in the opinion of the investigator, are unlikely to adhere to the requirements of the study or are unlikely to complete the vaccination and observation.
11. Subjects with any other finding which, in the opinion of the investigator or other delegated individual, would increase the risk of an adverse outcome from participation in the study.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited adverse events in children aged 4-11 years. | From the day of Dose 1 vaccination (Day 1) to 7 days post-Dose 1 vaccination
  Number and percentage of participants aged 4-11 years with solicited adverse events at the local injection site and systemically
Incidence of solicited adverse events in children aged 4-11 years. | From the day of Dose 2 vaccination (Day 56 days post-Dose 1) to 7 days post-Dose 2 vaccination
  Number and percentage of participants aged 4-11 years with solicited adverse events at the local injection site and systemically
Incidence of unsolicited serious adverse events | From the day of Dose 1 vaccination through 28 days post-Dose 2 vaccination (approximately 84 days)
  Number and percentage of participants with any untoward medical event
Vaccine-induced cellular immune responses to the Ebola virus glycoprotein (EBOV GP) | At Day 1 (Dose 1 vaccination)
  Proportion of participants with detectable EBOV-specific T cell subsets of interest
Vaccine-induced cellular immune responses to the Ebola virus glycoprotein (EBOV GP) | At Day 57 (56 days post-Dose 1 vaccination)
  Proportion of participants with detectable EBOV-specific T cell subsets of interest
Vaccine-induced cellular immune responses to the Ebola virus glycoprotein (EBOV GP) | At Day 78 (21 days post-Dose 2 vaccination)
  Proportion of participants with detectable EBOV-specific T cell subsets of interest

SECONDARY OUTCOMES:
Vaccine induced humoral immune responses to EBOV GP | At Day 1 (Dose 1 vaccination), Day 57 (56 days post-Dose 1 vaccination), and Day 78 (21 days post-Dose 2 vaccination)
  EBOV GP antibody concentration measured by ELISA

OTHER OUTCOMES:
Vaccine induced humoral immune response to EBOV GP | At Day 1 (Dose 1 vaccination), Day 57 (56 days post-Dose 1 vaccination), and Day 78 (21 days post-Dose 2 vaccination)
  EBOV GP antibody concentration measured by LUMINEX assay

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Watson-Jones, PhD, Study Chair — London School of Hygiene and Tropical Medicine
Locations (1):
- EBOVAC Kambia 1 clinic, Kambia, Sierra Leone

IPD SHARING:
Plan to Share IPD: Yes
The clinical trials results will be published in an open access, peer-reviewed journal, which will include, as feasible, the study protocol. A summary of the study results will be included within the trial resignation record in PACTR and ClinicalTrials.gov
Supporting Information: Study Protocol
Time Frame: within 12 months of the study completion date
Access Criteria: open